CLINICAL TRIAL: NCT01218087
Title: Cranial Cup Use for the Prevention of Positional Head Shape Deformity in the NICU
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study discontinued by DSMB due to loss of equipoise.
Sponsor: Boston Children's Hospital (Other)
Collaborators: Boston Orthotics & Prosthetics (Other)
Responsible Party: Principal Investigator, Michele DeGrazia, Director Nursing Research, NICU, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 08120584
Record Dates: First submitted 2010-09-30; First posted 2010-10-11 (Estimated); Results first posted 2015-08-26 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2016-12

CONDITIONS: Plagiocephaly; Scaphocephaly; Brachycephaly
Keywords: Positional Head Shape Deformity
MeSH Terms: conditions — Plagiocephaly; Craniosynostoses

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cranial cup device and Moldable positioner device (Experimental): The cranial cup for 12/24 hours and the moldable positioner device was used for positioning infants the remainder of the 24 hours
  Interventions: Device: Cranial cup device and Moldable positioner; Device: Moldable positioner device
- Moldable positioner device (Active Comparator): Moldable positioner device was used for positioning infants for 24/24 hours
  Interventions: Device: Moldable positioner device

INTERVENTIONS:
Device: Cranial cup device and Moldable positioner — The cranial cup device was used 12/24 hours (alternating with the moldable positioner device) and was evaluated for feasibility, safety and efficacy for preventing head shape deformity in hospitalized infants
  Arms: Cranial cup device and Moldable positioner device
Device: Moldable positioner device — This moldable positioning device was used 24/24 hours as a comparison to the cranial cup device.

SUMMARY:
Many hospitalized infants can develop a flattening of the back or sides of their head. This condition develops gradually when an infant's head rests on a firm or semi-firm surface for a prolonged period of time. Premature infants are more likely to have a positional head shape deformity because they may spend longer periods of time in a crib. Infants participating in this study will be randomly assigned to either standard treatment, which is a moldable positioner device, or to a cranial cup device and moldable positioner for positioning. The purpose of this prospective single-blinded randomized clinical trial will be to evaluate the effectiveness of the cranial cup in preventing positional head shape deformity in the NICU patient population.

DETAILED DESCRIPTION:
The primary outcome for this study will be cranial index and cranial symmetry measured at hospital discharge; the secondary outcome measure is the incidence of oxygen desaturation events (apnea, bradycardia and oxygen desaturation).

The pilot study was undertaken to evaluate if the cranial cup can be successfully incorporated into the NICU patient care regime, the pilot study included 5 infants.

The main trial enrollment was estimated to be 160 infants from 4 centers. Upon enrollment infants will be randomized to one of two study groups

* Cranial cup and moldable positioner
* Moldable positioner

Inclusion criteria:

There are several inclusion criteria for participation in the study:

1. Infants born at >/= 22 weeks gestation
2. Infant that are </= 7 days of age
3. Infants that receive medical clearance from their healthcare team
4. Infants that have an estimated minimum NICU length of stay = / > 14 days from the time of enrollment

Infants were stratified by study site and weight at enrollment (< 1000 grams versus = / > 1000 grams).

ELIGIBILITY:
Inclusion Criteria:

1. Infants born at >/= 22 weeks gestation
2. Infant that are </= 7 days of age
3. Infants that receive medical clearance from their healthcare team
4. Infants that have an estimated minimum NICU length of stay = / > 14 days from the time of enrollment

Exclusion Criteria:

1. Infants that require only prone positioning to maintain airway patency (such as those with Pierre Robin Syndrome/Sequence) will not be eligible to participate; this is because infants must be able to lie supine for at least part of the day to use the cranial cup
2. Infants requiring medical devices such as a continuous ventricular drain, subgaleal shunt, or intravenous catheters (unless placement of the IV is temporary) prevent proper positioning using the cranial cup
3. Infants with a craniofacial anomaly, cervical anomaly, or critical airway infants
4. Infants with Cutis Aplasia or significant skin breakdown to the scalp, because the cranial cup may worsen a preexisting condition
5. Infants with a prenatal diagnosis of craniosynostosis
6. Infants deemed not suitable for participation by the attending neonatologist
7. Infants that are to be transferred to a non-participating hospital within 14 days of enrollment as this timeframe may not be adequate to show a difference in head shapes

Max Age: 10 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2010-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele DeGrazia, PhD, NNP, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Approximately 800 infants from the 4 participating NICUs were screened; most were excluded for an anticipated length of stay of < 14 days, for medical reasons, and a few parents declined. The total number enrolled out of the approximately 800 screened was 88.
Groups:
- Cranial Cup Device: The cranial cup device was used 12/24 hours and the moldable positioner device was used for positioning infants the remainder of the 24 hours.
- Moldable Positioner Device: Moldable positioner device was used 24/24 hours as a comparison to the cranial cup and moldable positioner study arm.
Period: Overall Study
Arm/Group | Cranial Cup Device | Moldable Positioner Device
Started | 42 | 41
Completed | 27 | 35
Not Completed | 15 | 6
Not completed — Death | 2 | 1
Not completed — Withdrawal by Subject | 5 | 0
Not completed — Transferred | 8 | 5

BASELINE CHARACTERISTICS:
Population: Approximately 800 infants from the 4 participating NICUs were screened; most were excluded for an anticipated length of stay of < 14 days, for medical reasons, and a few parents declined. The total number enrolled out of the approximately 800 screened was 88.
Groups:
- Cranial Cup Device: cranial cup device: The cranial cup device was used 12/24 hours (alternating with the moldable positioner device) and was evaluated for feasibility, safety and efficacy for preventing head shape deformity in the infant
- Moldable Positioner Device: moldable positioner device: This positioning device was used 24/24 hours as a comparison to the cranial cup device.
- Total: Total of all reporting groups
Arm/Group | Cranial Cup Device | Moldable Positioner Device | Total
Number analyzed (Participants) | 27 | 35 | 62
Age, Continuous [Median (Full Range); unit: days] | 0 [0 to 7] | 0 [0 to 12] | 0 [0 to 12]
Gender [Count of Participants; unit: Participants]
  Female | 9 | 13 | 22
  Male | 18 | 22 | 40
Race/Ethnicity, Customized [Number; unit: participants]
  White | 15 | 26 | 41
  African American | 7 | 7 | 14
  Asian | 1 | 0 | 1
  Native Hawaiian | 0 | 1 | 1
  Hispanic | 4 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 27 | 35 | 62

OUTCOME MEASURES:

1. Primary Outcome: Cranial Abnormalities Were Measured at Hospital Discharge
Description: Cranial abnormality measurements were obtained at hospital discharge by orthotists blinded to the study group assignment. Cranial abnormalities include both cranial index measures and cranial symmetry measures. Cranial index (normal measurement between 73%-85%) was obtained dividing the head width (M-L) by length (A-P) then multiplying it by 100%. Cranial symmetry (normal measurement of<8mm) was obtained by calculating the difference in the right and left anterior-posterior measures.
Time Frame: up to 120 days
Measure: Number; unit: % participant cranial abnormalities
Groups:
- Cranial Cup Device: cranial cup device: The cranial cup device was used 12/24 hours (alternating with the moldable positioner device) and was evaluated for feasibility, safety and efficacy for preventing head shape deformity in the infant. Although infants in this arm did use the moldable positioner, they were analyzed separately from the comparison group.
Arm/Group | Cranial Cup Device | Moldable Positioner Device
Number analyzed (Participants) | 27 | 35
% participant cranial abnormalities | 46 | 19
Statistical Analysis 1: Comparison: Cranial Cup Device vs Moldable Positioner Device; Test type: Non-Inferiority or Equivalence — Following the first interim analysis of the first 40 infants, the sample size calculation was revised. A revised sample size of 62 infants (31 per treatment arm) was based on an observed reduction of 41% to 11% in the experimental group with a goal p value of 0.01; p = 0.03, Fisher Exact

2. Secondary Outcome: Incidence of Cardiorespiratory
Description: daily log of cardiorespiratory events (apnea, bradycardia, oxygen desaturation) collected on a daily positioning log at the infant's bedside
Time Frame: daily up to 120 days
Measure: Number; unit: cardioresp. events/100hrs of device use
Arm/Group | Cranial Cup Device | Moldable Positioner Device
Number analyzed (Participants) | 27 | 35
cardioresp. events/100hrs of device use | 5.4 | 5.9

ADVERSE EVENTS:
Arm/Group | Cranial Cup Device | Moldable Positioner Device
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/35
Other Adverse Events (participants affected / at risk) | 0/27 | 0/35

LIMITATIONS AND CAVEATS:
During the second interim analysis, safety monitors recommended early closure due to loss of study equipoise. Clinical staff had been reporting observable differences in infant head shapes for the two study groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes